CLINICAL TRIAL: NCT02301793
Title: Educating Nurses About Venous Thromboembolism Prevention
Brief Title: Educating Nurses About Venous Thromboembolism (VTE) Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NA_00043860
Record Dates: First submitted 2014-11-22; First posted 2014-11-26 (Estimated); Results first posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Venous Thromboembolism; Venous Thrombosis
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis

STUDY DESIGN:
Intervention Model Description: One arm was provided linear static education (Static) using PowerPoint slides with voiceover to cover the concepts. The other arm was provided interactive learner-centric dynamic scenario-based education (Dynamic), where each scenario resulted in either positive reinforcement or corrective feedback with an opportunity to apply knowledge to a new scenario.
Who Masked: Participant, Outcomes Assessor
Masking Description: Within strata, a coin toss (ERH) was used to randomize floors into either the Dynamic education arm or the Static education arm. Based on the outcome of the coin toss, nurses were then remotely assigned the online education module by an institutional nurse educator (DLS). The assigned educational module then appeared in the nurse's list of education assignments for completion within the institutional Learning Management System. Nurses are required to complete clinically relevant education regularly as part of ongoing professional practice and a waiver of consent was provided by the IRB; therefore nurses were not aware of their participation in a trial nor were they aware that two education modules existed. Additionally, the VTE prophylaxis medication non-administration dataset provided to the biostatistical team (i.e. outcomes assessors) for analysis was blinded by treatment arm and department.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contemporary Education Format (Experimental): Nurses in this arm received education about venous thromboembolism (VTE) in a web-based contemporary interactive format.
  Intervention: Nurse education in contemporary format
  Interventions: Behavioral: Nurse education in contemporary format
- Traditional Education Format (Active Comparator): Nurses in this arm received education about venous thromboembolism (VTE) in a web-based traditional linear PowerPoint format with voice over.
  Intervention: Nurse education in traditional format
  Interventions: Behavioral: Nurse education in traditional format

INTERVENTIONS:
Behavioral: Nurse education in contemporary format — Education about VTE was delivered through a web-based contemporary interactive format
  Arms: Contemporary Education Format
Behavioral: Nurse education in traditional format — Education about VTE was delivered through a web-based traditional linear Powerpoint format with voice over.
  Arms: Traditional Education Format

SUMMARY:
As part of mandatory on-going nursing education, the investigators have incorporated identical information into two distinct web-based learning formats - the traditional linear PowerPoint format (with voice-over) and a new interactive format developed with central nursing education.

The investigators will cluster randomize nurses by floor to receive either the traditional education or the new interactive education, and evaluate the impact on administration of VTE prophylaxis doses administered by nurses before and after education. All nurses on a floor will receive the same educational format. If one method of education results in statistically significant improvement in VTE prophylaxis administration, the investigators will cross over to deliver the superior education format to all nurses who originally were given the less effective method.

DETAILED DESCRIPTION:
BACKGROUND

* In an attempt to improve venous thromboembolism (VTE) prophylaxis adherence the investigators carried out qualitative studies to obtain patients' viewpoints on how nurses should be educated about VTE prevention and to assess nurses' beliefs and perceptions about pharmacologic VTE prophylaxis
* The investigators observed deficiencies in nurses' knowledge and misconceptions about VTE prophylaxis that likely lowers adherence to administration of prescribed VTE prophylaxis doses
* As a part of our original Patient-Centered Outcomes Research Institute (PCORI) proposal, the investigators planned to educate nurses to address the observed deficiencies and misconceptions and improve their ability to communicate effectively with patients

  * Historically, nurse education has been done via a linear, PowerPoint-based platform with voice-over but with no interactive component (TRADITIONAL)
  * A newer platform for nurse education became available for use and includes scenario-based teaching, ongoing assessment, and immediate remediation. Most importantly, it is a highly interactive product (CONTEMPORARY)

STUDY DESIGN AND ANALYTIC PLAN

* Research hypotheses

  * Primary: Nurse participants who receive either of these interventions will improve administration of prescribed VTE prophylaxis evidenced by a decrease in frequency of non-administered doses of VTE prophylaxis, compared with their frequency at baseline.
  * Secondary: Nurse participants who receive the contemporary education format will have a larger decrease in frequency of missed doses of VTE prophylaxis compared with those who participate in the traditional education format.
* Study Design

  * Cluster Randomized Trial 21 floors, block randomized by floor type (medicine [n=11] vs. surgery [n=10]) and (ICU [n=5] vs. non-ICU [n=16]) All nurses on each floor are assigned the same education type to mitigate issues related to contamination if nurses discuss the education with their colleagues
* Primary Outcome measure: Proportion of non-administered doses of pharmacological VTE prophylaxis (dose level)
* Secondary Outcome Measures:

  * Proportion of doses documented as missed due to patient refusal (dose level)
  * Proportion of patients with any VTE (patient level)
  * Proportion of patients with Deep Vein Thrombosis (DVT) (patient level)
  * Proportion of patients with Pulmonary Embolism (PE) (patient level)
* Analytic methods

  * Primary analyses - Intention-to-treat (includes all nurses assigned, whether or not they completed the education) Is there a difference between units allocated to either of the interventions comparing their outcome measure to their baseline measure? Is there a difference comparing those who received the contemporary education format vs. the traditional education format?
  * Secondary analysis - Per protocol (includes only nurses who completed the education) Do nurses who receive education perform better (improved administration of prescribed VTE prophylaxis) than those who did not? Do nurses who received the education in the contemporary format perform better than those who received it in the traditional format

ELIGIBILITY:
Inclusion Criteria:

* Nurses on selected surgical and medical floors at Johns Hopkins Hospital

Exclusion Criteria:

* Nurses who were not permanently associated with one of the 21 hospital floors (e.g. traveling nurse, float nurse) were excluded from this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 933 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2015-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliott R Haut, MD PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shermock KM, Lau BD, Haut ER, Hobson DB, Ganetsky VS, Kraus PS, Efird LE, Lehmann CU, Pinto BL, Ross PA, Streiff MB. Patterns of non-administration of ordered doses of venous thromboembolism prophylaxis: implications for novel intervention strategies. PLoS One. 2013 Jun 14;8(6):e66311. doi: 10.1371/journal.pone.0066311. Print 2013. PMID 23799091
- [Background] Elder S, Hobson DB, Rand CS, Streiff MB, Haut ER, Efird LE, Kraus PS, Lehmann CU, Shermock KM. Hidden Barriers to Delivery of Pharmacological Venous Thromboembolism Prophylaxis: The Role of Nursing Beliefs and Practices. J Patient Saf. 2016 Jun;12(2):63-8. doi: 10.1097/PTS.0000000000000086. PMID 24681420
- [Derived] Lau BD, Shaffer DL, Hobson DB, Yenokyan G, Wang J, Sugar EA, Canner JK, Bongiovanni D, Kraus PS, Popoola VO, Shihab HM, Farrow NE, Aboagye JK, Pronovost PJ, Streiff MB, Haut ER. Effectiveness of two distinct web-based education tools for bedside nurses on medication administration practice for venous thromboembolism prevention: A randomized clinical trial. PLoS One. 2017 Aug 16;12(8):e0181664. doi: 10.1371/journal.pone.0181664. eCollection 2017. PMID 28813425
- See also: PCORI Website Page - "Improving Patient-Nurse Communication to Prevent a Life-Threatening Complication" — http://www.pcori.org/research-in-action/improving-patient-nurse-communication-prevent-life-threatening-complication
- See also: PCORI Website Page - "Preventing Venous Thromboembolism: Empowering Patients and Enabling Patient-Centered Care via Health Information Technology" — http://www.pcori.org/research-results/2013/preventing-venous-thromboembolism-empowering-patients-and-enabling-patient
- See also: Website to take the nurse education module. "Venous Thromboembolism Prevention: The Nurse's Perspective" — https://www.hopkinsmedicine.org/armstrong_institute/improvement_projects/infections_complications/VTE/strategies.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nurses were identified using our centralized education directory that associates nurses with their designated departments and hospital floors. On July 23, 2014, nurses were cluster randomized by floor to receive one of two education modules about VTE prevention. Nurses were asked to complete their assigned education module by October 23, 2014.
Pre-assignment Details: Pre Education Study Period reflects the baseline participants information (patient visits). Post Education Study Period reflects the participants information following the implementation of the nurse education intervention.
Units Other Than Participants: Patient visits
Groups:
- Contemporary Education Format: Nurses in this arm received education about venous thromboembolism (VTE) in a web-based contemporary interactive format.
  Intervention: Nurse education in contemporary format
  Nurse education in contemporary format: Education about VTE was delivered through a web-based contemporary interactive format
- Traditional Education Format: Nurses in this arm received education about venous thromboembolism (VTE) in a web-based traditional linear PowerPoint format with voice over.
  Intervention: Nurse education in traditional format
  Nurse education in traditional format: Education about VTE was delivered through a web-based traditional linear Powerpoint format with voice over.
Period: Pre Education Study Period
Arm/Group | Contemporary Education Format | Traditional Education Format
Started | NA; 2722 Patient visits (Nurses had not been randomized) | NA; 2603 Patient visits (Nurses had not been randomized)
Completed | NA; 2722 Patient visits (Nurses had not been randomized) | NA; 2603 Patient visits (Nurses had not been randomized)
Not Completed | NA; 0 Patient visits | NA; 0 Patient visits
Period: During and Post Education Study Period
Arm/Group | Contemporary Education Format | Traditional Education Format
Started | 488; 6566 Patient visits | 445; 5355 Patient visits
Completed | 405; 6566 Patient visits | 396; 5355 Patient visits
Not Completed | 83; 0 Patient visits | 49; 0 Patient visits

BASELINE CHARACTERISTICS:
Population: Outcomes assessed were analyzed on patient visit level as each encounter represents a unique participant outcome. Patient A might receive all doses during their first visit and miss doses during a second visit. Patient A might have been in different Arms during different visits. Baseline information was only collected during the pre-education phase
Units Other Than Participants: Patient Visit
Groups:
- Total: Total of all reporting groups
Arm/Group | Contemporary Education Format | Traditional Education Format | Total
Number analyzed (Participants) | 1925 | 2021 | 3946
Number analyzed (Patient Visit) | 2722 | 2603 | 5325
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (16.9) | 56.3 (17.3) | 56 (17.1)
Sex: Female, Male [Count of Units; unit: Patient Visit] — Population: The numbers of patients were 2,722 and 2603, in the dynamic and static groups respectively. While the unique number of patients were 1925, and 2021 respectively.
  Patient Visit
    Female | 1435 | 1186 | 2621
    Male | 1287 | 1417 | 2704
Race (NIH/OMB) [Count of Units; unit: Patient Visit]
  American Indian or Alaska Native | 4 | 7 | 11
  Asian | 46 | 50 | 96
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1106 | 980 | 2086
  White | 1367 | 1396 | 2763
  More than one race | 199 | 170 | 369
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Patient Visit]
  United States | 2722 | 2603 | 5325

OUTCOME MEASURES:

1. Primary Outcome: Non Administration of Prescribed VTE Prophylaxis Medication Doses
Description: This is the percentage of VTE prophylaxis doses that were not administered for any reason as documented in the electronic health record by a nurse
Time Frame: (Baseline); approximately 3 months later (Post-Education)
Population: The total number of patient visits in each study arm. Overall number of participants represents the number of unique patients in the study. These numbers reflect patient visits at baseline and following the implementation of the nurse education intervention.
Measure: Number (95% Confidence Interval); unit: percentage of nonadministration
Units Other Than Participants: patient visits
Arm/Group | Contemporary Education Format | Traditional Education Format
Number analyzed (Participants) | 4686 | 4398
Number analyzed (patient visits) | 6835 | 5941
percentage of nonadministration
  Pre-Education: number analyzed (Participants) | 1925 | 2021
  Pre-Education: number analyzed (patient visits) | 2722 | 2603
  Pre-Education | 10.8 [7.7 to 15.0] | 14.5 [10.2 to 20.4]
  Post-Education: number analyzed (Participants) | 2761 | 2377
  Post-Education: number analyzed (patient visits) | 4113 | 3338
  Post-Education | 9.2 [6.6 to 12.8] | 13.5 [9.6 to 19.1]
Statistical Analysis 1: Comparison: Contemporary Education Format vs Traditional Education Format; The hypothesis comparing the different educational arms was evaluated using an intention-to-treat approach (i.e. all nurses were included regardless of training completion) accounting for clustering in the data and comparing rates of VTE prophylaxis dose non-administration at baseline and during the Post-Education period. Two per-protocol sensitivity analyses were performed. They compared the Baseline vs. Post-Education periods for nurses who received training and nurses who completed training; Test type: Other; p = 0.05, Regression, Logistic — The reported p-values were calculated by reiterating the multiple outputation procedure 1000 times, we estimated the odds ratios (ORs) and their 95% confidence intervals conditional on the floor and nurse; Odds Ratio (OR) = 1

2. Secondary Outcome: Rates of All VTE Among Hospitalized Patients
Description: Did the intervention decrease rates of VTE among hospitalized patients?
Time Frame: 3-12 months after end of study
Population: Data were not collected
Arm/Group | Contemporary Education Format | Traditional Education Format
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Rates of Deep Vein Thrombosis (DVT) Among Hospitalized Patients
Description: Did the intervention decrease rates of DVT among hospitalized patients?
Time Frame: 3-12 months after end of study
Population: Data were not collected
Arm/Group | Contemporary Education Format | Traditional Education Format
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Rates of Pulmonary Embolism (PE) Among Hospitalized Patients
Description: Did the intervention decrease rates of PE among hospitalized patients?
Time Frame: 3-12 months after end of study
Population: Data were not collected
Arm/Group | Contemporary Education Format | Traditional Education Format
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Proportion of Non Administration of Prescribed VTE Prophylaxis Medication Doses Which Are Documented as Patient Refusal
Description: Did the intervention decrease rates of patient refusal of VTE prophylaxis medication doses among hospitalized patients?
Time Frame: Baseline; approximately 3 months later (post education)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patient refused doses
Units Other Than Participants: patient visits
Arm/Group | Contemporary Education Format | Traditional Education Format
Number analyzed (Participants) | 4686 | 4398
Number analyzed (patient visits) | 6835 | 5941
percentage of patient refused doses
  Pre-Education: number analyzed (Participants) | 1925 | 2021
  Pre-Education: number analyzed (patient visits) | 2722 | 2603
  Pre-Education | 5.6 [3.1 to 10.0] | 7.3 [4.0 to 13.2]
  Post-Education: number analyzed (Participants) | 2761 | 2377
  Post-Education: number analyzed (patient visits) | 4113 | 3338
  Post-Education | 5.1 [2.8 to 9.0] | 7.0 [3.8 to 12.6]
Statistical Analysis 1: Comparison: Contemporary Education Format vs Traditional Education Format; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.05, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events were reported at patient visit level
Arm/Group | Contemporary Education Format | Traditional Education Format
All-Cause Mortality (participants affected / at risk) | 0/6835 | 0/5941
Serious Adverse Events (participants affected / at risk) | 0/6835 | 0/5941
Other Adverse Events (participants affected / at risk) | 0/6835 | 0/5941

LIMITATIONS AND CAVEATS:
This trial was conducted in a single center potentially limiting the generalizability of our findings. The differences associated with education by specific clinical department in the current study was not explored.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT02301793/Prot_SAP_000.pdf